CLINICAL TRIAL: NCT02239094
Title: Identification of Biosignatures for Lurasidone (Latuda) Response in Bipolar Depression
Brief Title: Biosignatures of Latuda for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6954; 6954 (Other: NYSPI IRB)
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Bipolar Depression
Keywords: Bipolar Disorder; depression; Bipolar depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone (Latuda) (Other): All study participants will receive open-label Latuda.
  Interventions: Drug: Lurasidone (Latuda)

INTERVENTIONS:
Drug: Lurasidone (Latuda) — Antipsychotic medication approved for use with Bipolar disorder
  Other Names: Latuda

SUMMARY:
The study proposes to conduct a pilot study of biological predictors of lurasidone response in bipolar depression.

DETAILED DESCRIPTION:
The study proposes to enroll 20 participants with a bipolar disorder who are currently in an episode of major depression.Magnetic resonance imaging (MRI), recordings of brain electrical activity (EEG), and psychological testing to explore possible predictors of lurasidone treatment response will be conducted. Blood samples will be collected for a future study of blood protein predictors of response. After testing, participants will receive an open-label 8-week trial of lurasidone (Latuda™) at approved dosage levels. Participants who attain remission of their major depressive episode will be eligible for a six-month continuation phase to explore predictors of sustained response to continuation treatment. Data analyses will use statistical testing to explore potential biological predictors of lurasidone response. This will provide a framework for clarifying which patients are best suited to this treatment and begin to develop a model for precision treatment of this difficult-to-treat disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 60
2. Outpatients with a primary Diagnostic and Statistical Manual of the American Psychiatric Association, Fourth Edition (DSM-IV) diagnosis of Bipolar Disorder I, II, or NOS (Not Otherwise Specified)
3. Current episode of Major Depression
4. At least moderate severity of depression
5. Agrees to, and is eligible for, electroencephalogram (EEG) / psychological testing, magnetic resonance imaging (MRI), and blood draws
6. Provides informed consent

Exclusion Criteria:

1. Current drug or alcohol abuse/dependence, except nicotine (within 6 months for dependence; 2 for abuse)
2. Taking any of the following exclusionary medications: antipsychotics, anticonvulsants, mood stabilizers, stimulants, antidepressant medications, medications with significant interactions with lurasidone, except during the washout prior to testing and blood collection
3. Unstable medical condition, including significant liver disease, hypothyroidism (i.e., condition not adequately stabilized for 3 months), and conditions likely to require hospitalization or with a life expectancy of < 6 mos.*
4. Patients considered at significant risk for suicide
5. Inadequate understanding of English
6. Currently pregnant or breast-feeding; fecund women not using adequate contraceptive methods; plan to become pregnant within 12 months
7. Contraindications to MRI (e.g. ferromagnetic body implants, history of metal working, etc.)
8. Have epilepsy, neuromuscular disorder, or tardive dyskinesia
9. Require immediate hospitalization for psychiatric disorder
10. Require medications for a general medical condition that contraindicate any study medication**
11. Receiving or have received during the index episode vagus nerve stimulation, electroconvulsive therapy, transcranial magnetic stimulation, or other somatic treatments
12. Allergy to, or other medical contraindication to lurasidone treatment
13. Currently enrolled in another research study, and participation in that study contraindicates participation
14. Clinically significant screening laboratory abnormalities (* see below)
15. Currently taking an effective mood stabilizer and/or antidepressant regimen
16. Inability to undergo a three week medication-free period, including history of significant clinical deterioration from past periods off medication or when medication dosage was reduced, including mania, severe depression, etc.
17. Any reason not listed herein that would make participation in the study hazardous *Medical criteria for exclusion:

    * Untreated hypertension: > 140/90 Torr on repeated measurement (If hypertension becomes stabilized, subject may enroll in study)
    * Hepatitis: any liver function test > 2x the upper limit of normal
    * Renal failure: estimated Glomerular Filtration Rate (eGFR, corrected for body surface area) repeatedly < 30 mL/min
    * Hypothyroidism: thryrotropin stimulating hormone level > upper limit of normal (unless accompanied by other euthyroid indices and the confirmation by an internist or endocrinologist that this does not represent hypothyroidism)
    * Anemia: hemoglobin < 10 grams/deciliter (borderline hemoglobin must be of known origin, stable, and not clinically significant)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Lan MJ, Pantazatos SP, Ogden RT, Rubin-Falcone H, Hellerstein D, McGrath PJ, Mann JJ. Resting State MRI Amplitude of Low Frequency Fluctuations Associated With Suicidal Ideation in Bipolar Depression. J Clin Psychiatry. 2022 Mar 30;83(3):21m14054. doi: 10.4088/JCP.21m14054. PMID 35377567
- See also: Depression Evaluation Service (site location) website — http://www.depression-nyc.org
- See also: Institutional department website — http://columbiapsychiatry.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone (Latuda)
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Remitted before started | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone (Latuda)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Rating Scale for Depression (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression.
  Nine of the items are based upon patient report, and one is on the rater's observation during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone (Latuda)
Number analyzed (Participants) | 18
units on a scale | 24.3 (6.4)

2. Primary Outcome: Montgomery-Asberg Rating Scale for Depression (MADRS) at Week8
Description: as for outcome 1
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone (Latuda)
Number analyzed (Participants) | 18
units on a scale | 8 (8.2)

ADVERSE EVENTS:
Time Frame: Adverse event was carefully monitored throughout the whole study period (8 Weeks)
Arm/Group | Lurasidone (Latuda)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 8/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (Latuda) (N=18)
Headache (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (5)
Weight Gain (Metabolism and nutrition disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
No healthy volunteer group and no placebo comparisons. And this is an open label treatment study.The results are also limited by the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No